CLINICAL TRIAL: NCT02752282
Title: Anticipatory Counseling on LNG-IUS Continuation, Utilization and Satisfaction
Acronym: ACCCUSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Bayer (Industry); Cook County Health (Other Government); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Emily Godfrey, Associate Professor, Family Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 49648
Record Dates: First submitted 2016-04-15; First posted 2016-04-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Vaginal Bleeding; Uterine Cramping
Keywords: Family Planning; LNG-IUS; Health Education
MeSH Terms: conditions — Uterine Hemorrhage; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Video (Sham Comparator): Participants in this study arm will be assigned to watch a short educational video about new pap screening guidelines for women. Intervention: Cancer Screening Guidelines.
  Interventions: Other: Cancer Screening Guidelines
- Intervention Video (Active Comparator): Participants in this group will be assigned to watch a short educational video providing anticipatory counseling on their LNG-IUS' side effects and expected changes in bleeding. Intervention: Anticipatory Counseling
  Interventions: Other: Anticipatory Counseling

INTERVENTIONS:
Other: Anticipatory Counseling — Anticipatory Counseling provides information on expected side-effects that may change or go away over time, or stay for the duration of the treatment. Anticipatory counseling can also help patients understand when their side-effects are normal and when to seek medical attention.
  Arms: Intervention Video
Other: Cancer Screening Guidelines — Anticipatory Counseling on United States Preventative Services Task Force (USPSTF) updated pap screening guidelines
  Arms: Control Video

SUMMARY:
This study is a counseling intervention for new LNG-IUS users. The study explores the use of video technology to deliver anticipatory counseling on LNG-IUS side-effects, adjustment periods and bleeding changes to women newly using the LNG-IUS for contraceptive purposes. The primary aim is to understand if anticipatory counseling delivered via video can increase LNG-IUS satisfaction and continuation of the device in the first 6 months of use.

DETAILED DESCRIPTION:
Enhanced anticipatory counseling detailing side effects when initiating progestin-only injectable contraception improved its continued use among women.While continuation rates at one year among levonorgestrel intrauterine system (LNG-IUS) users are considerably higher than those for progestin-only injectable users in the United States (80% versus 56%), enhanced anticipatory counseling could have an impact on the 20% of LNG IUS users who choose to discontinue the method within one year of use. For this reason, the investigators propose a study that would develop and pilot-test an anticipatory counseling intervention detailing unscheduled bleeding and other side effects such as pelvic pain or cramping among new LNG IUS users and compare this with a "control," using video technology. The investigators have chosen video technology for the counseling intervention to ensure that all participants receive the exact same information about LNG side effects, which would be not possible using a face-to-face clinician-participant counseling model.

The investigators propose three phases for this study. In Phase 1, a systematic literature search evaluating effective components in videos used for contraceptive counseling and the development of two separate video scripts will lead to: (1) an intervention, detailing expected side effects and safety of the LNG IUS, and (2) a similar-looking "control," detailing only recommended screening guidelines for women, as well as information about LNG IUS safety. This phase of the study uses focus groups prior to the development of the video interventions, initially with family planning experts for content accuracy and cultural sensitivity, and secondarily with new LNG IUS users for acceptability. Findings from this phase will be used to fine-tune the scripts prior to the development of the videos.

In Phase 2 of the study, the investigators will pilot a trial in the clinical setting to evaluate the anticipatory counseling video intervention and its impact on LNG-IUS knowledge, continuation, health care utilization, and satisfaction. After receiving comprehensive contraceptive counseling from their clinicians, women who choose to have the LNG IUS inserted will be given a brochure that asks them to participate in an online study. After signing-on to an innovative website, participants will be randomized to either an intervention or control video and complete short questionnaires related to demographics, baseline menstruation, satisfaction, and LNG IUS knowledge before and after viewing their assigned video. Women will be followed for six months. They will be asked to complete a short online survey at three and six months regarding LNG IUS continuation, health care utilization, and satisfaction. Findings from this study will serve to design a future, appropriately powered randomized controlled trial assessing LNG IUS continuation, utilization, and satisfaction rates at 12 months.

In Phase 3, we will use the findings from Phase 2 to develop a similar protocol and recruit up to 178 women at three sites across the US to test the same primary aims of the video: LNG-IUS continuation, utilization, and satisfaction over a 12 month period. In phase 3, subjects will be randomized to watch either the control or intervention video.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 and over who are deemed appropriate candidates be their healthcare providers and choose to use LNG-IUS, either Mirena or Skyla.
2. Within five days of FIRST using either Mirena or Skyla
3. Willing to answer online questions before and after watching the assigned video (intervention or control)
4. Willing to complete short online questionnaire at three and six months
5. Has working email and/or phone number
6. Able to understand verbal and written English
7. Appropriate LNG-IUS candidates whoa re being treated for other pre-existing medical disorders while using the LNG IUS may continue to take their medications as directed by their healthcare provider.

Exclusion Criteria:

1. Women aged less than 18 years old
2. Initiated LNG-IUS method more than five days from enrollment date.
3. Within six weeks postpartum
4. Breastfeeding
5. Using LNG-IUS for treatment other than contraception
6. Do not have access to the Web
7. Have neither working email or phone number
8. Does not understand written or verbal English
9. Inappropriate candidates for LNG IUS as deemed by healthcare provider

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in LNG-IUS knowledge, satisfaction and continuation from baseline | 6 months
  Using standardize questionnaires we will assess any significant differences in LNG-IUS knowledge, satisfaction or continuation after 6 months between control arm and intervention arm subjects.

SECONDARY OUTCOMES:
Percent of subjects in Phase II who complete all 3 surveys on-time over 6 months compared by recruitment method and site | 6 months
  Assess what percent of study participants were successfully recruited via a brochure or email contact at Seattle and Chicago.
Number of subjects reporting LNG-IUS discontinuation during the study time frame (6 months) by reason for LNG-IUS removal | 6 months
  Track number of subjects who have their LNG-IUS removed during the study period by reason, including: bleeding, cramping, acne, weight gain, depression or other reasons.
LNG-IUS user self-reported satisfaction with video counseling | 6 months
  A survey using modified likert scales and free text boxes, will ask participants how helpful the video was, how many times they watched the video, and any feedback they had about video elements to improve.
LNG-IUS user self-reported LNG-IUS healthcare utilization during study period | baseline, 3 months, 6 months
  Compare LNG-IUS user self-reported healthcare utilization at baseline (before the LNg-IUS was placed) with 3 and 6 months after LNG-IUS use. This include number of phone calls and office visits and the user reported helpfulness of these interactions with their healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Godfrey, MD, MPH, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Stroger Hospital of Cook County, Chicago, Illinois
  - University of Washington Medical Centers, Seattle, Washington